CLINICAL TRIAL: NCT01474967
Title: Effect of Dosage of Metformin on Menstruation and Lipid Profile in Women With Polycystic Ovary Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hormozgan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Hamidreza Mahboobi, Resident, Hormozgan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Metformin in PCOS
Record Dates: First submitted 2011-11-16; First posted 2011-11-18 (Estimated); Last update posted 2011-11-21 (Estimated); Status verified 2011-11

CONDITIONS: Polycystic Ovary Syndrome
Keywords: polycystic ovary syndrome; lipid profile; metformin
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lower metformin dose group (Experimental): 500 mg metformin daily with breakfast for 1 week 500 mg metformin per 12 hours with breakfast and dinner for 23 weeks
  Interventions: Drug: Metformin
- Higher metformin dose group (Active Comparator): 500 mg metfomin daily with breakfast for 1 week 500 mg metformin per 12 hours with breakfast and dinner for 1 week 500 mg metformin with breakfast and 1000 mg with dinner for 22 weeks
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — 500 mg metformin daily with breakfast for 1 week 500 mg metformin per 12 hours with breakfast and dinner for 1 week 500 mg metformin with breakfast and 1000 mg with dinner for 22 weeks
  Other Names: metformex
  Arms: Higher metformin dose group
Drug: Metformin — 500 mg metfomin daily with breakfast for 1 week 500 mg metformin per 12 hours with breakfast and dinner for 23 weeks
  Other Names: metformex
  Arms: Lower metformin dose group

SUMMARY:
Polycystic ovarian syndrome (PCOS) is the most common cause of anovulatory infertility and causes menstrual disruption in 6.6-6.8% of women in reproductive age and is characterized by insulin resistance, hyperinsulinemia, hyperandrogenism and anovulation. The gaol of this study was to assess the effects of metformin on menstrual disorders and lipid profile in women with PCOS in bandarabbas.

DETAILED DESCRIPTION:
Poly cystic ovarian syndrome (PCOS) is a common hormonal disorder in women that affecting of 6.6-6.8% of women o f reproductive age. PCOS associated with a broad range of clinical, hormonal and metabolic disorders consist of hirsutism, Obesity, Acne and elevated male hormones, anovulatory cycles, dyslipidemia and infertility.

Metformin is an oral hyperglycemic agent witch by decrease insulin resistance and improving serum glucose level in diabetic patients and anovulatory cyle in women with PCOS. The goal of this study is to evaluate the efficacy of different dosage of metformin on menstruation and lipid profile in women with PCOS in banda-abbas.

ELIGIBILITY:
Inclusion Criteria:

* Women with PCOS

Exclusion Criteria:

* avoiding to participate in the study

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-02; Primary Completion 2011-01 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Lipid profile | 6 month
  The serum levels of Cholesterol, LDL, HDL and Triglyceride were measured before and after of treatment in both groups.

SECONDARY OUTCOMES:
Hormone levels | 6 month
  LH, FSH, Testosterone

CONTACTS AND LOCATIONS:
Overall Officials: Nazanin Abdi, resident, Principal Investigator — Hormozgan University of Medical Sciences (HUMS)
Locations (1):
- Hormozgan University of Medical Sciences (HUMS), Bandarabbas, Hormozgan, Iran